CLINICAL TRIAL: NCT04253210
Title: Body Positive Images and Photo Modification Cues on Social Media
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study plans did not materialize due to the COVID-19 pandemic.
Sponsor: Chapman University (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-20-42
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Body Image

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sexualized images / High photo modification (Experimental)
  Interventions: Other: psychological
- Sexualized images / Low photo modification (Experimental)
  Interventions: Other: psychological
- Nonsexualized images / High photo modification (Experimental)
  Interventions: Other: psychological
- Nonsexualized images / Low photo modification (Experimental)
  Interventions: Other: psychological
- Control images (Experimental)
  Interventions: Other: psychological

INTERVENTIONS:
Other: psychological — Participants will either view body positive images that are sexualized (vs. nonsexualized) and a great deal of evidence of photo modification (vs. low photo modification).

SUMMARY:
The purpose of this research is to explore how women evaluate photos of other women posted on social media sites. There are two factors the investigators plan to explore in an online experiment: (a) the degree to which body positive images appear to be sexualized or not; and (b) whether or not there is evidence of photo modification on these images. The results of this work will provide greater understanding into the effects of the body positive movement and determine conditions under which these campaigns are most impactful.

DETAILED DESCRIPTION:
The purpose of this research is to explore how women evaluate photos of other women posted on social media sites. Specifically, the investigators are interested in providing more nuance regarding the effectiveness of body positive imagery (i.e., more diverse representations of physical attractiveness and empowerment of women underrepresented in the mainstream media). The literature on female objectification suggests women are oftentimes portrayed in unrealistic ways (e.g., ultra-thin and hyper-sexualized) via the mainstream media. Moreover, warranting theory provides predictions about the extent to which online content represents an offline reality. As such, there are two factors the investigators plan to explore in an online experiment: (a) the degree to which body positive images appear to be sexualized or not; and (b) whether or not there is evidence of photo modification on these images. The results of this work will provide greater understanding into the effects of the body positive movement and determine conditions under which these campaigns are most impactful.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Closed-Ended Questionnaire Items Extent of Sexualization (semantic differential) | During the single-session study (data collected over 12 months); immediately after viewing experimental images
  Closed-Ended Questionnaire Items--Participants will be asked to report to what extent they believe the images that they viewed are sexual in nature using semantic differential scales.
Closed-Ended Questionnaire Items Extent of Physical Attractiveness (semantic differential) | During the single-session study (data collected over 12 months); immediately after viewing experimental images
  Closed-Ended Questionnaire Items--Participants will be asked to report to what extent they believe the people in the images that they viewed are attractive using a semantic differential scale.
Closed-Ended Questionnaire Items of Extent of Photo Modification (Likert Scale) | During the single-session study (data collected over 12 months); immediately after viewing experimental images
  Closed-Ended Questionnaire Items--Participants will be asked to report to what extent they believe the images that they viewed were modified or edited in some way with a series of statements about photo modification (1 = strongly disagree; 7 = strongly agree).
Closed-Ended Questionnaire Items of Extent of Body Appreciation | During the single-session study (data collected over 12 months); immediately after viewing experimental images
  Closed-Ended Questionnaire Items--Participants will be asked to report to what extent they feel appreciative of their own body with a series of statements about body appreciation (1 = strongly disagree; 7 = strongly agree).
Closed-Ended Questionnaire Items of Extent of Positive Body Image (Likert Scale) | During the single-session study (data collected over 12 months); immediately after viewing experimental images
  Closed-Ended Questionnaire Items--Participants will be asked to report about their feelings about their own body a series of statements on their body (1 = strongly disagree; 7 = strongly agree).
Closed-Ended Questionnaire Items of Extent of Positive Evaluations of Photos (Likert Scale) | During the single-session study (data collected over 12 months); immediately after viewing experimental images
  Closed-Ended Questionnaire Items--Participants will be asked to report their evaluations of the images that they viewed on Likert scales with a series of statements (1 = strongly disagree; 7 = strongly agree).
Open-Ended Questionnaire Items on the Rate of Other-Objectification / Social Aggression | During the single-session study (data collected over 12 months); as they view the experimental images
  Open-Ended Questionnaire Items--Participants will be asked to report their feelings about the images they are viewing in open-ended response boxes to assess the extent to which they objectify and/or express social aggression toward the images.
Open-Ended Questionnaire Items on the Rate of State Self-Objectification | During the single-session study (data collected over 12 months); immediately after viewing experimental images
  Open-Ended Questionnaire Items--Participants will be asked to report 20 statements about themselves and their identity in open-ended response boxes.
Closed-Ended Demographic Item of Biological Sex | During the single-session study (data collected over 12 months); at the end of the survey with other demographic measures
  Questionnaire Item--Participants will report their biological sex as "male" or "female" to include in sample characteristics.
Closed-Ended Demographic Item of Race/Ethnicity | During the single-session study (data collected over 12 months); at the end of the survey with other demographic measures
  Questionnaire Item--Participants will report their race/ethnic background" to include in sample characteristics.
Closed-Ended Demographic Item of Age | During the single-session study (data collected over 12 months); at the end of the survey with other demographic measures
  Questionnaire Item--Participants will report their age to include in sample characteristics.
Closed-Ended Demographic Item of Social Media Use | During the single-session study (data collected over 12 months); at the end of the survey with other demographic measures
  Questionnaire Item--Participants will report wether they have an Instagram account ("yes" or "no"); if "yes," they will be asked to indicate how much time per day they spend on Instagram.
Closed-Ended Demographic Item of Body Height | During the single-session study (data collected over 12 months); at the end of the survey with other demographic measures
  Questionnaire Item--Participants will report their height (feet/inches) to include in sample characteristics.
Closed-Ended Demographic Item of Body Weight | During the single-session study (data collected over 12 months); at the end of the survey with other demographic measures
  Questionnaire Item--Participants will report their weight (in pounds) to include in sample characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Chapman University, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided